CLINICAL TRIAL: NCT01618266
Title: Study of Ozurdex® Treatment Practice in Patients With Macular Oedema Due to Retinal Vein Occlusion
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: MAF/AGN/OPH/RET/009
Record Dates: First submitted 2012-06-11; First posted 2012-06-13 (Estimated); Results first posted 2016-02-11 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-02

CONDITIONS: Macular Edema; Retinal Vein Occlusion
MeSH Terms: conditions — Macular Edema; Retinal Vein Occlusion | interventions — Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ozurdex® (dexamethasone intravitreal implant): dexamethasone intravitreal implant 700 μg administered into the eye according to physician judgment.
  Interventions: Drug: dexamethasone intravitreal implant

INTERVENTIONS:
Drug: dexamethasone intravitreal implant — dexamethasone intravitreal implant 700 μg administered into the eye according to physician judgment.
  Other Names: Ozurdex®

SUMMARY:
Epidemiological study of Ozurdex® in sites treating patients with retinal vein occlusion.

ELIGIBILITY:
Inclusion Criteria:

* Macular oedema due to retinal vein occlusion

Exclusion Criteria:

* Not living in metropolitan France

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Macular Oedema due to Retinal Vein Occlusion
Sampling Method: Non-Probability Sample
Enrollment: 375 (Actual)
Dates: Start 2011-11; Primary Completion 2013-04 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Paris, France

REFERENCES:
- [Derived] Korobelnik JF, Kodjikian L, Delcourt C, Gualino V, Leaback R, Pinchinat S, Velard ME. Two-year, prospective, multicenter study of the use of dexamethasone intravitreal implant for treatment of macular edema secondary to retinal vein occlusion in the clinical setting in France. Graefes Arch Clin Exp Ophthalmol. 2016 Dec;254(12):2307-2318. doi: 10.1007/s00417-016-3394-y. Epub 2016 Jun 11. PMID 27286894

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ozurdex® (Dexamethasone Intravitreal Implant)
Started | 375
Completed | 279
Not Completed | 96
Not completed — Lost to Follow-up | 9
Not completed — Treatment satisfaction | 10
Not completed — Other reasons | 11
Not completed — Lack of Efficacy | 23
Not completed — Protocol Violation | 43

BASELINE CHARACTERISTICS:
Arm/Group | Ozurdex® (Dexamethasone Intravitreal Implant)
Number analyzed (Participants) | 375
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.31 (11.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 169
  Male | 206

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA) in the Study Eye
Description: BCVA is measured in the study eye using an eye chart and is reported as the number of letters read correctly (ranging from 0 to 100 letters). The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). The higher the number of letters read correctly, the better the vision (or visual acuity). A positive number change in the number of letters read means that the vision improved and a negative number change in the number of letters read means that the vision has worsened.
Time Frame: Baseline, Month 6
Population: All enrolled patients
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Ozurdex® (Dexamethasone Intravitreal Implant)
Number analyzed (Participants) | 375
Letters
  Baseline | 47.56 (21.21)
  Change from Baseline at Month 6 (N=323) | 5.09 (19.02)

2. Secondary Outcome: Change From Baseline in BCVA in the Study Eye Diagnosed With Branch Retinal Vein Occlusion (BRVO)
Description: BCVA is measured in the study eye using an eye chart and is reported as the number of letters read correctly (ranging from 0 to 100 letters). The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). The higher the number of letters read correctly, the better the vision (or visual acuity). A positive number change in the number of letters read means that the vision improved and a negative number change in the number of letters read means that the vision has worsened. BRVO is a blockage of the small veins in the retina.
Time Frame: Baseline, Month 6
Population: All enrolled patients with BRVO
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Ozurdex® (Dexamethasone Intravitreal Implant)
Number analyzed (Participants) | 202
Letters
  Baseline | 52.80 (17.42)
  Change from Baseline at Month 6 | 5.50 (19.59)

3. Secondary Outcome: Change From Baseline in BCVA in the Study Eye Diagnosed With Central Retinal Vein Occlusion (CRVO)
Description: BCVA is measured in the study eye using an eye chart and is reported as the number of letters read correctly (ranging from 0 to 100 letters). The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). The higher the number of letters read correctly, the better the vision (or visual acuity). A positive number change in the number of letters read means that the vision improved and a negative number change in the number of letters read means that the vision has worsened. CRVO is a blockage of the main vein in the retina.
Time Frame: Baseline, Month 6
Population: All enrolled patients with CRVO
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Ozurdex® (Dexamethasone Intravitreal Implant)
Number analyzed (Participants) | 173
Letters
  Baseline | 41.45 (23.54)
  Change from Baseline at Month 6 | 4.63 (18.38)

4. Secondary Outcome: Change From Baseline in BCVA in the Study Eye in Previously Treatment Naïve Patients
Description: BCVA is measured in the study eye using an eye chart and is reported as the number of letters read correctly (ranging from 0 to 100 letters). The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). The higher the number of letters read correctly, the better the vision (or visual acuity). A positive number change in the number of letters read means that the vision improved and a negative number change in the number of letters read means that the vision has worsened. Treatment naïve patients have not been previously treated for retinal vein occlusion.
Time Frame: Baseline, Month 6
Population: All enrolled patients who were treatment naïve
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Ozurdex® (Dexamethasone Intravitreal Implant)
Number analyzed (Participants) | 145
Letters
  Baseline | 43.94 (23.12)
  Change from Baseline at Month 6 | 7.45 (20.00)

5. Secondary Outcome: Change From Baseline in BCVA in the Study Eye in Patients Previously Treated With Ozurdex®
Description: BCVA is measured in the study eye using an eye chart and is reported as the number of letters read correctly (ranging from 0 to 100 letters). The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). The higher the number of letters read correctly, the better the vision (or visual acuity). A positive number change in the number of letters read means that the vision improved and a negative number change in the number of letters read means that the vision has worsened. Previous treatment for retinal vein occlusion was Ozurdex®.
Time Frame: Baseline, Month 6
Population: All enrolled patients previously treated with Ozurdex®
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Ozurdex® (Dexamethasone Intravitreal Implant)
Number analyzed (Participants) | 149
Letters
  Baseline | 52.46 (18.90)
  Change from Baseline at Month 6 | 1.95 (16.03)

6. Secondary Outcome: Change From Baseline in BCVA in the Study Eye in Patients Previously Naïve to Ozurdex® Treatment
Description: BCVA is measured in the study eye using an eye chart and is reported as the number of letters read correctly (ranging from 0 to 100 letters). The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). The higher the number of letters read correctly, the better the vision (or visual acuity). A positive number change in the number of letters read means that the vision improved and a negative number change in the number of letters read means that the vision has worsened. Patients naive to Ozurdex® have not been previously treated for retinal vein occlusion.
Time Frame: Baseline, Month 6
Population: All enrolled patients previously naïve to Ozurdex® treatment
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Ozurdex® (Dexamethasone Intravitreal Implant)
Number analyzed (Participants) | 79
Letters
  Baseline | 45.29 (20.20)
  Change from Baseline at Month 6 | 8.39 (21.10)

7. Secondary Outcome: Change From Baseline in BCVA in the Study Eye Based on Macular Edema Onset <3 Months
Description: BCVA is measured in the study eye using an eye chart and is reported as the number of letters read correctly (ranging from 0 to 100 letters). The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). The higher the number of letters read correctly, the better the vision (or visual acuity). A positive number change in the number of letters read means that the vision improved and a negative number change in the number of letters read means that the vision has worsened. The onset of macular edema was <3 months prior to treatment.
Time Frame: Baseline, Month 6
Population: All enrolled patients with macular edema onset <3 months
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Ozurdex® (Dexamethasone Intravitreal Implant)
Number analyzed (Participants) | 180
Letters
  Baseline | 43.27 (22.83)
  Change from Baseline at Month 6 | 8.53 (20.50)

8. Secondary Outcome: Change From Baseline in BCVA in the Study Eye Based on Macular Edema Onset ≥3 Months
Description: BCVA is measured in the study eye using an eye chart and is reported as the number of letters read correctly (ranging from 0 to 100 letters). The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). The higher the number of letters read correctly, the better the vision (or visual acuity). A positive number change in the number of letters read means that the vision improved and a negative number change in the number of letters read means that the vision has worsened. The onset of macular edema was ≥3 months prior to treatment.
Time Frame: Baseline, Month 6
Population: All enrolled patients with macular edema onset ≥3 months
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Ozurdex® (Dexamethasone Intravitreal Implant)
Number analyzed (Participants) | 183
Letters
  Baseline | 51.44 (19.00)
  Change from Baseline at Month 6 | 1.96 (17.47)

9. Secondary Outcome: Change From Baseline in BCVA in the Study Eye in Patients Only Treated With Ozurdex®
Description: BCVA is measured in the study eye using an eye chart and is reported as the number of letters read correctly (ranging from 0 to 100 letters). The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). The higher the number of letters read correctly, the better the vision (or visual acuity). A positive number change in the number of letters read means that the vision improved and a negative number change in the number of letters read means that the vision has worsened. Patients had only been previously treated with Ozurdex®.
Time Frame: Baseline, Month 6
Population: All enrolled patients only treated with Ozurdex
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Ozurdex® (Dexamethasone Intravitreal Implant)
Number analyzed (Participants) | 254
Letters
  Baseline | 49.28 (19.23)
  Change from Baseline at Month 6 | 5.48 (18.77)

10. Secondary Outcome: Change From Baseline in BCVA in the Study Eye in Patients Receiving Ozurdex® and Then Other RVO Treatments
Description: BCVA is measured in the study eye using an eye chart and is reported as the number of letters read correctly (ranging from 0 to 100 letters). The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). The higher the number of letters read correctly, the better the vision (or visual acuity). A positive number change in the number of letters read means that the vision improved and a negative number change in the number of letters read means that the vision has worsened. Patients were previously treated with Ozurdex® and then switched to other RVO treatment during the study.
Time Frame: Baseline, Month 6
Population: All enrolled patients receiving Ozurdex® and then other RVO treatments
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Ozurdex® (Dexamethasone Intravitreal Implant)
Number analyzed (Participants) | 121
Letters
  Baseline | 43.97 (24.57)
  Change from Baseline at Month 6 | 4.25 (19.61)

11. Secondary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA) in the Study Eye
Description: as for outcome 1
Time Frame: Baseline, Week 6, Month 4, Month 12, Month 18, Month 24
Population: All enrolled patients
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Ozurdex® (Dexamethasone Intravitreal Implant)
Number analyzed (Participants) | 375
Letters
  Baseline | 47.6 (21.2)
  Change from Baseline at Week 6 (N=350) | 11.41 (16.4)
  Change from Baseline at Month 4 (N=337) | 3.08 (18.2)
  Change from Baseline at Month 12 (N=306) | 2.85 (21.4)
  Change from Baseline at Month 18 (N=287) | 3.02 (22.2)
  Change from Baseline at Month 24 (N=274) | 4.64 (22.3)

12. Secondary Outcome: Percentage of Patients With BCVA Improvement of ≥15 Letters From Baseline in the Study Eye
Description: BCVA is measured in the study eye using an eye chart and is reported as the number of letters read correctly (ranging from 0 to 100 letters). The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). The higher the number of letters read correctly, the better the vision (or visual acuity). An increase in the number of letters read correctly indicates improvement and a decrease in the number of letters read correctly indicates a worsening.
Time Frame: Baseline, Month 24
Population: All enrolled patients
Measure: Number; unit: Percentage of Patients
Arm/Group | Ozurdex® (Dexamethasone Intravitreal Implant)
Number analyzed (Participants) | 375
Percentage of Patients | 38.7

ADVERSE EVENTS:
Arm/Group | Ozurdex® (Dexamethasone Intravitreal Implant)
Serious Adverse Events (participants affected / at risk) | 98/375
Other Adverse Events (participants affected / at risk) | 252/375
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Ozurdex® (Dexamethasone Intravitreal Implant) (N=375)
Ocular Hypertension (Eye disorders) | 32
Cataract (Eye disorders) | 26
Glaucoma (Eye disorders) | 6
Cataract Surgery (Surgical and medical procedures) | 3
Vitreous Haemorrhage (Eye disorders) | 3
Stroke (Nervous system disorders) | 2
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2
Macular Fibrosis (Eye disorders) | 2
Death (General disorders) | 2
Cardiac Arrest (Cardiac disorders) | 1
Subscapular Cataract (Eye disorders) | 1
Sudden Falls Due to Legs Giving Way (Nervous system disorders) | 1
Diabetes (Metabolism and nutrition disorders) | 1
Detached Retina (Eye disorders) | 1
Cardiopulmonary Arrest (Cardiac disorders) | 1
Macular Degeneration (Eye disorders) | 1
Hypertension (Vascular disorders) | 1
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1/206 — MALES ONLY
Infarction (Vascular disorders) | 1
Pulmonary Infection (Infections and infestations) | 1
Retinal Ischaemia (Eye disorders) | 1
Herpetic Keratitis (Infections and infestations) | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Acute Pancreatitis (Gastrointestinal disorders) | 1
Coronary Artery Bypass (Surgical and medical procedures) | 1
Pulmonary Arterial Thrombosis (Vascular disorders) | 1
Pulmonary Disorder (Respiratory, thoracic and mediastinal disorders) | 1
Prostate tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/206 — MALES ONLY
Transient Ischaemic Attack (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ozurdex® (Dexamethasone Intravitreal Implant) (N=375)
Ocular Hypertension (Eye disorders) | 128
Cataract (Eye disorders) | 124

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.